CLINICAL TRIAL: NCT05191368
Title: Yunnan University of Traditional Chinese Medicine
Brief Title: Safety and Immunogenicity of Sars-cov-2 Vaccine in Patients With Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yunnan University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ting Zhao, doctor, Yunnan University of Chinese Medicine
Other Study IDs: Yunnan University of CM
Record Dates: First submitted 2022-01-12; First posted 2022-01-13 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Rheumatic Disease
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal group: Healthy people who received two doses of COVID-19 vaccine
  Interventions: Other: No intervention
- RA Patients injected with 2 doses of vaccine: RA Patients who received two doses of COVID-19 vaccine
  Interventions: Other: No intervention
- Unvaccinated RA patients: RA Patients who received zero doses of COVID-19 vaccine
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study was to preliminarily evaluate the immunogenicity of sars-cov-2 vaccine in patients with rheumatic diseases. The clinical information collection and blood sample testing of 100 healthy people and 200 patients with rheumatic diseases will be completed in Yunnan Traditional Chinese medicine hospital.

Research methods and procedures: clinical information collection and blood sample detection were carried out in healthy people and patients with rheumatic diseases, including systemic lupus erythematosus (SLE), antiphospholipid syndrome (APS), rheumatoid arthritis (RA), Sjogren's syndrome (SS), systemic sclerosis (SSC), idiopathic inflammatory myopathy (IIM), systemic vasculitis and spinal arthritis

DETAILED DESCRIPTION:
Rheumatic diseases (RDS) are a large class of systemic diseases caused by genetic background, environment and physics, infection, metabolism, endocrine, immune response and other reasons, mainly involving joints and surrounding tissues. The diseases covered include systemic lupus erythematosus (SLE), antiphospholipid syndrome (APS), rheumatoid arthritis (RA) Sjogren's syndrome (SS), systemic sclerosis (SSC), idiopathic inflammatory myopathy (IIM), systemic vasculitis, spinal arthritis, etc. Patients with rheumatic diseases have an increased risk of infection due to autoimmune dysfunction and long-term use of hormones and immunosuppressants.

The incidence rate of coronary heart disease (COVID-19) pandemic caused by severe acute respiratory syndrome coronavirus 2 (severe acute respiratory syndrome coronavirus 2, SARS-CoV-2) in 2019 has resulted in high incidence and mortality worldwide. Although the epidemic prevention measures such as keeping distance and quarantine isolation have effectively improved and limited the epidemic scope and the number of infected people, the groups with low immunity are still the susceptible groups of sars-cov-2.

Vaccination is very important to suppress the epidemic and reduce the overall mortality. It can protect people from sars-cov-2 infection and the deterioration of covid-192, and has good safety. However, there are not enough reports on the safety and immunogenicity of sars-cov-2 vaccine in patients with rheumatic diseases. Studies have reported that the immunogenicity of sars-cov-2 vaccine is reduced in immunocompromised patients, including the use of immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of rheumatic diseases in western medicine;

  * 18-70 years old, male or female;

    * The patient voluntarily participated in this clinical study, has been informed of relevant matters, and signed the informed consent form

Exclusion Criteria:

It does not meet the diagnostic criteria of rheumatic diseases in western medicine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ① Meet the diagnostic criteria of rheumatic diseases in western medicine;
  ② 18-70 years old, male or female;
  ③ The patient voluntarily participated in this clinical study, has been informed of relevant matters, and signed the informed consent form
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Sars-cov-2 neutralizing antibody | 2022.01.01
  Inhibition rate of sars-cov-2 neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Fanying Meng, Study Director — Yunnan University of Chinese Medicine
Locations (1):
- Yunnan University of traditional Chinese Medicine, Kunming, Kunming, China

IPD SHARING:
Plan to Share IPD: No